CLINICAL TRIAL: NCT01420146
Title: Pilot Imaging Study With 89Zr-Trastuzumab in HER2-positive Metastatic Breast Cancer Patients : Correlation With FDG-PET/CT and Anatomopathological Results
Brief Title: Pilot Imaging Study With 89Zr-Trastuzumab in HER2-positive Metastatic Breast Cancer Patients
Acronym: IJBMNZrT003
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IJBMNZrT003
Record Dates: First submitted 2011-08-08; First posted 2011-08-19 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2015-01

CONDITIONS: Breast Neoplasms; Secondary; HER2 Positive Carcinoma of Breast
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zr89-trastuzumab PET/CT (Experimental): Zr89-trastuzumab PET/CT single arm
  Interventions: Drug: Zr89-trastuzumab

INTERVENTIONS:
Drug: Zr89-trastuzumab — trastuzumab labelled with zirconium 89 for PET/CT
  Other Names: HER2 ImmunoPET/CT; HER2 receptor imaging; Breast cancer molecular imaging

SUMMARY:
Evaluation of the diagnostic potential of HER2 imaging using zirconium 89 labelled trastuzumab.

DETAILED DESCRIPTION:
This is the first belgian feasibility study of HER2 imaging using a labelled monoclonal antibody, namely trastuzumab labelled with zirconium 89.

The aims of this study are:

I/ Evaluate the diagnostic potential of HER2 imaging using zirconium 89 labelled trastuzumab (based on the Groningen experience), through the analysis of the correlation between the FDG-PET/CT and the HER2 immunoPET.

II/ PET quantification of HER2 receptor by using the images and the blood pharmacokinetic of the tracer.

III/ In the subset of patients for whom biopsies of metastatic sites have not been carried out previously and are of an easy access, tissue will be acquired as part of the validation of the HER2 immunoPET and as an attempt to better understand the molecular heterogeneity of HER2 positive breast cancer at the time of relapse.

IV/Evaluate the concentration of circulating HER2 extracellular domain in the blood and study his possible role as on imaging quality

ELIGIBILITY:
Inclusion criteria:

1. All patients selected for this imaging study are patients scheduled to start trastuzumab-based therapy for advanced HER2 positive breast cancer (This includes trastuzumab alone, trastuzumab + chemotherapy, trastuzumab + endocrine therapy).
2. Histologically confirmed HER 2 positive (defined as FISH amplification ratio more than 2.2) invasive carcinoma of the breast (primary tumor at diagnosis) with locally recurrent or metastatic disease.
3. Patients with FDG-PET positive metastatic lesions.
4. Brain metastases are allowed provided they are controlled and they are not the sole site of metastatic disease.
5. Patient planned to have metastatic site biopsy for HER2 status control.
6. Age ≥ 18 years
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 to 1
8. For women of childbearing potential a pregnancy test will be done and an agreement to use a highly-effective non hormonal form of contraception.
9. Agreement from the patient to participate in this imaging study and if indicated agreement to biopsy one or two accessible lesions.
10. Signed written informed consent (approved by the Ethics Committee) obtained prior to any study procedure

Exclusion criteria:

1. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)
2. Pregnant or lactating women
3. Current known infection with HIV, HBV, or HCV
4. Known severe hypersensitivity to trastuzumab
5. Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol
6. Patients with bone only metastases are not eligible
7. Psychiatric illness/social situations that would limit compliance with study requirements
8. Patients who received lapatinib within the 7 days prior to HER immunoPET/CT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Flamen, MD, PhD, Principal Investigator — Jules Bordet Institut
Locations (1):
- Jules Bordet Institut, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Zr89-trastuzumab PET/CT: Zr89-trastuzumab (trastuzumab labelled with zirconium 89) for PET/CT single arm
Period: Overall Study
Arm/Group | Zr89-trastuzumab PET/CT
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Zr89-trastuzumab PET/CT
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 20

OUTCOME MEASURES:

1. Primary Outcome: Test the Diagnostic Accuracy of the HER2 Imaging Using the Labelled Monoclonal Antibody Trastuzumab by Correlating the HER2 PET/CT Imaging With the FDG-PET/CT and Molecular Characterization of Tumor Samples With Discordant Image Findings
Description: A visual 'patient-based' classification capturing the whole disease burden was developed by using a side-by-side display, comparing baseline FDG-PET/CT(showing all FDG-positive mets independent of their HER2-imaging status) & day4 HER2-PET/CT. Pts were grouped into 4 HER2-PET/CT patterns according to the proportion of FDG avid tumour load showing relevant 89Zr-T uptake. Pattern A: entire tumor load showed pertinent tracer uptake; B: dominant part of tumour load showed tracer uptake; C: minor part of tumor load showed tracer uptake; D: entire tumor load lacked tracer uptake. Patterns A+B='HER2-positive' & C+D='HER2-negative'. In the 20 pts: 4 pts were classified "A", 5"B", 1"C" & 10"D". This classification indicates substantial heterogeneity of 89Zr-T uptake within this so called 'HER2-positive' pt population. After dichotomization, 11(55%) pts were considered as HER2-PET/CT negative. Furthermore, HER2-PET/CT revealed intrapatient heterogeneity of tumour uptake(pts classified B or C).
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Zr89-trastuzumab PET/CT
Number analyzed (Participants) | 20
Participants
  Pattern A | 4
  Pattern B | 5
  Pattern C | 1
  Pattern D | 10

2. Secondary Outcome: Time Activity Curve
Description: Time activity curve of normal organ and tumor lesions: pharmacokinetic
Time Frame: blood sample at 5, 15, 30, 60 minutes, 1 day, 2 days and 4 or 6 days after tracer injection. Images : Day 0, Day 2 and Day 4 or 6
Reporting Status: Not Posted

3. Secondary Outcome: HER2 Extracellular Domain
Description: evaluate the concentration of circulating HER2 extracellular domain in the blood and study his possible role as on imaging quality
Time Frame: within 60 min before tracer injection
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Zr89-trastuzumab PET/CT
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 10/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zr89-trastuzumab PET/CT (N=20)
Nausea - Pyrexia - Myalgia (General disorders) | 1 (3) — one SAE case containing 3 single events: * Gastrointestinal disorders : Nausea * General disorders and administration site conditions: Pyrexia * Musculoskeletal and connective tissue disorders: Myalgia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zr89-trastuzumab PET/CT (N=20)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Chills (General disorders) | 4 (4)
Hypersensitivity (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Pyrexia (General disorders) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes